CLINICAL TRIAL: NCT06787937
Title: Communicating About Nicotine and Differential Risks of Tobacco Products in Priority Populations
Brief Title: Communicating About Nicotine Reduction in Cigarettes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Emory University (Other); University of South Carolina (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lyudmila Popova, Associate Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H25318; R01CA239308 (NIH)
Record Dates: First submitted 2024-12-25; First posted 2025-01-22 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Tobacco Products; Smoking Behavior; Cigarette Use
Keywords: smoking; health communication; very low nicotine cigarettes
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VLNC with message campaign (Experimental): Participants in this arm will receive VLNCs during weekly visits and be exposed to messaging about VLNCs and reduced nicotine policy through multiple formats, including inserts placed in cigarette packs, printed advertisements, and videos presented during weekly visits.
  Interventions: Behavioral: VLNC messages
- VLNC only (Other): Participants in this arm will receive VLNCs during weekly visits but will not receive any messaging related to cigarettes or reduced nicotine policy. Instead, they will only be exposed to control messages, such as advertisements for bottled water, during weekly visits.
  Interventions: Behavioral: Control message

INTERVENTIONS:
Behavioral: VLNC messages — Participants will be exposed to messaging about VLNCs and reduced nicotine policy through multiple formats, including inserts placed in cigarette packs, printed advertisements, and video materials presented during their weekly visits.
  Arms: VLNC with message campaign
Behavioral: Control message — Participants will be exposed to control messages, such as advertisements for bottled water, during their weekly visits.
  Arms: VLNC only

SUMMARY:
The goal of this clinical trial is to learn how a messaging campaign about reduced nicotine cigarettes and policy, combined with the use of very low nicotine cigarettes (VLNCs), affects smoking behavior and attitudes among adult smokers. The study also aims to assess the efficacy of the messages in different populations, including smokers with past-month serious psychological distress (SPD), low socioeconomic status (SES), and those in neither category.

The primary hypothesis is: exposure to messages in combination with VLNC use will lead to less cigarettes use compared to VLNCs without messages.

Researchers will compare: The effects of receiving VLNCs with messages (treatment group) to receiving VLNCs without messages (control group).

Participants will: Complete a baseline survey and be randomly assigned to one of two groups: treatment (VLNCs + messages) or control (VLNCs only). Attend weekly study visits for surveys, breath samples, and receive supply of VLNCs , either with or without the messaging campaign. Complete brief daily surveys through text messages.

DETAILED DESCRIPTION:
This is a randomized, open label, controlled, two-site study to test the efficacy of a messaging campaign about reduced nicotine cigarettes and policy in combination with the use of very low nicotine cigarettes (VLNCs). Smokers from three groups: with past-month serious psychological distress (SPD), with low socioeconomic status (SES), and in neither category will complete a 1-week baseline and a 4-week study; they will be randomized to one of two conditions:

1. treatment condition, where participants receive VLNCs during weekly visits and are exposed to messages about VLNCs and reduced nicotine policy.
2. control condition, where participants receive VLNCs without exposure to messages.

Message intervention: Messages about VLNCs and reduced nicotine policy will be professionally developed as full-color inserts (small leaflets that will be inserted into cigarette packs given to participants), print ads, and videos. At each weekly visit, participants will see 3-6 messages about VLNCs and reduced nicotine policy (in the treatment condition) or, in the control condition, 3-6 messages unrelated to tobacco (ads for bottled water, which are neutral messages that are unlikely to affect tobacco-related perceptions or behavior). Participants in the treatment conditions will also have inserts in their VLNC cigarette packs.

Baseline visit: Participants will complete a baseline survey, provide expired breath Carbon Monoxide (CO) sample, and receive a 1-week supply of the study cigarettes (full nicotine).

Randomization visit: Participants will be randomized into either the treatment (VLNCs + messages) or control (VLNCs only) condition. Participants will complete questionnaires, provide an expired CO sample, and receive a 14-day supply of VLNCs (either with or without the messages, according to the assigned condition).

Weekly visits: Starting one week after the randomization visit, participants will complete 4 weekly visits at their designated study site. At each visit, they will complete questionnaires, provide an expired CO sample, and receive a 14-day supply of VLNCs (with or without the messages, according to the assigned condition).

Daily logs: Throughout the baseline and 4 weekly study periods, participants will receive daily text messages with links to brief online surveys.

ELIGIBILITY:
Inclusion Criteria:

* Age 21+ years
* Current smoker (self-report as having smoked 100 cigarettes in their lifetime and currently smoking on 27+ days out of past 30, expired breath carbon monoxide [CO] ≥6ppm to assess regular smoking)
* Can speak, read, and write in English
* Available for period of study
* Willing to try novel research cigarettes

Exclusion Criteria:

* Pregnancy or lactation
* Member of the same household as a study subject
* Unwilling to use research cigarettes as part of the trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1230 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Cigarettes per day | Week 4 of the trial (post randomization)
  Number of cigarettes smoked per day (study and non-study cigarettes).
  * Averaged number of cigarettes smoked based on 7 days' daily logs submitted through text-based survey during the last week of the trial.
  * Response: integer indicating number per day.

SECONDARY OUTCOMES:
Use of other tobacco products | Week 4 of the trial (post randomization)
  Amount of other combusted (LCCs) and noncombustible (e-cigarettes) products per day.
  * Averaged number of other tobacco products is based on 7 days' daily logs submitted through text-based survey during the last week of the trial.
  * Response: integer indicating number per day.
Use of cessation medications | Week 4 of the trial (post randomization)
  Use of nicotine replacement therapy or prescription cessation medications in the past 24 hours based on 7 days' daily logs submitted through text-based survey during the last week of the trial. This will be assessed using a multiple-choice question, allowing participants to select all NRT or prescription cessation medications used from a provided list of options.
Forgoing cigarettes | Through study completion, up to 4 weeks
  One item measures number of times forgoing cigarettes when considering smoking in the past 24 hours based on daily logs submitted through text-based survey from baseline visit to the end of the trial. Response options are: 1 (Never), 2 (Once), 3 (A few times), and 4 (Lots of times), with higher scores representing a better outcome.
Making a quit attempt | Through study completion, up to 4 weeks
  One item measures whether participants have made an attempt to stop smoking (not smoking cigarettes for at least 24 hours) in the past week based on questionnaire completed at weekly in-person visits throughout the trial. Response options: 1 (yes), 2 (no), 3 (don't know).
Perceived risk of smoking VLNCs | Week 4 of the trial (post randomization)
  One item measures perceived likelihood of overall harm to health under conditions of smoking VLNCs based on questionnaire completed at the week 4 visit. Response options range from 1 (Not at all likely) to 5 (Extremely likely), with higher scores representing a better outcome. An additional option, "Don't know", is also provided.
Self-efficacy to quit | Week 4 of the trial (post randomization)
  Multiple items assess perceptions about strength of confidence in own ability to quit smoking based on questionnaire completed at week 4 visit. Response options range from 1 (not at all) to 7 (extremely), with higher scores representing a better outcome. An additional option, "Don't know", is also provided.
Intention to quit smoking | Week 4 of the trial (post randomization)
  Multiple items assesses Intentions and motivation to quit smoking in the next month and 6 months based on questionnaire completed at week 4 visit. Response options range from 1 (not at all) to 7 (extremely), with higher scores representing a better outcome. An additional option, "Don't know", is also provided.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Georgia State university, Atlanta, Georgia
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pei D, Juris A, Nkansah P, Thrasher JF, Giordano NA, Henderson KC, Spears CA, Ashley DL, Mallory VC, Adeniji FP, Foster JD, Ni W, Kodriati N, Ogunnaike A, Pechacek TF, Kirpich A, Popova L. Nicotine Intervention and Communication for Empowering Reduction (NICER): study protocol for a randomized controlled trial among priority populations of people who smoke. Trials. 2025 Nov 17;26(1):514. doi: 10.1186/s13063-025-09216-8. PMID 41250122